CLINICAL TRIAL: NCT02511782
Title: Use of a Transdermal Patch to Noninvasively Monitor Inflammatory Biomarkers of Acute and Chronic Skin GVHD
Brief Title: Transdermal Patch to Monitor Inflammatory Biomarkers of GVHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-0212
Record Dates: First submitted 2015-06-10; First posted 2015-07-30 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Graft Versus Host Disease
Keywords: children; bone marrow transplant; GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acute Graft versus Host Disease (Experimental): This study arm includes patients who undergo allogeneic hematopoietic cell transplantation at CCHMC and develop acute graft versus host disease. Skin cell samples will be collected using the D-SQUAME Skin Sampling Discs. The first baseline skin sample will be obtained prior to the preparative regimen for stem cell transplant. Samples will be collected weekly after stem cell infusion until 8 weeks, if acute GVHD does not develop. If acute GVHD does develop, weekly samples will continue to be collected until resolution of acute GVHD or development of chronic GVHD, whichever occurs first. Blood samples will be collected at these same time points.
  Interventions: Device: D-SQUAME Skin Sampling Discs
- Chronic Graft versus Host Disease (Experimental): This study arm includes patients who undergo allogeneic hematopoietic cell transplantation at CCHMC and develop chronic graft versus host disease. Skin cell samples will be collected weekly for 4 weeks using the D-SQUAME Skin Sampling Discs. Blood samples will be collected at these same time points.
  Interventions: Device: D-SQUAME Skin Sampling Discs
- Healthy Controls (Active Comparator): This study arm includes healthy age matched controls as comparisons to study participants who develop graft versus host disease. These controls may be either healthy age matched siblings of patients who develop acute graft versus host disease or healthy age matched siblings of patients that are seen in the bone marrow transplant, oncology, or hematology clinics. A one-time single skin cell sample will be collected using a D-SQUAME Skin Sampling Disc. Blood samples will not be collected from the healthy controls.
  Interventions: Device: D-SQUAME Skin Sampling Discs

INTERVENTIONS:
Device: D-SQUAME Skin Sampling Discs — A D-SQUAME Skin Sampling Disc is a noninvasive patch that collects skin cell samples when affixed to the superficial stratum corneum (top layer of skin). The patch is applied with gentle pressure to the desired quadrant of the forearm and removed 2 minutes after application.

SUMMARY:
The aim of this study is to measure local inflammatory responses in patients undergoing an allogeneic stem cell transplant and attempt to define any set of biomarkers that are significantly altered in acute or chronic skin graft versus host disease.

DETAILED DESCRIPTION:
Acute skin graft versus host disease is a significant complication following allogeneic stem cell transplant. To date, there are no specific dermal biomarkers that predict or define the onset of acute skin graft versus host disease. The primary objective of this study is to observe the changes in the inflammatory environment of the skin during the process of acute and chronic skin graft versus host disease. This will be accomplished by using a non-invasive transdermal patch called D-Squame to analyze inflammatory cytokines and key epidermal proteins. Patients will be enrolled prior to receiving a stem cell transplant and followed weekly after stem cell infusion until day 99. If acute skin graft versus host disease develops, they will be followed weekly until resolution of acute graft versus host disease or development of chronic graft versus host disease, whichever occurs first. Patients with a diagnosis of chronic skin graft versus host disease will be enrolled and followed weekly until 4 weeks, irrespective of clinical course. In addition, healthy controls will be enrolled and used as comparators. The relevance of this study is to provide a better understanding of the local inflammatory environment induced by acute or chronic skin graft versus host disease. This is likely to enable the investigators to define a biomarker panel that predicts the onset of acute graft versus host disease rapidly and non-invasively.

ELIGIBILITY:
Inclusion criteria for patients who may develop acute graft versus host disease:

* All patients undergoing an allogeneic hematopoietic stem cell transplant at CCHMC.
* All conditioning regimens are eligible.

Exclusion criteria for patients who may develop acute graft versus host disease:

• Pre-existing skin conditions like, but not limited to epidermolysis bullosa, psoriasis, acne, or cellulitis.

Inclusion criteria for patients who have chronic graft versus host disease:

* Bone marrow transplant performed at CCHMC or an outside institution.
* Diagnosis of chronic skin graft versus host disease.

Exclusion criteria for patients who have chronic graft versus host disease:

• Bone marrow transplant performed for epidermolysis bullosa.

Inclusion criteria for controls:

* Healthy volunteers.
* Age matched to the patients with existing acute skin graft versus host disease.

Exclusion criteria for controls:

• Pre-existing dermatologic conditions. (E.g. eczema, psoriasis, acne etc.)

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Graft Versus Host Disease | Chronic Graft Versus Host Disease | Healthy Controls
Started | 51 | 2 | 10
Completed | 50 | 2 | 10
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Graft Versus Host Disease | Chronic Graft Versus Host Disease | Healthy Controls | Total
Number analyzed (Participants) | 51 | 2 | 10 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51 | 2 | 10 | 63
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 0 | 5 | 21
  Male | 35 | 2 | 5 | 42

OUTCOME MEASURES:

1. Primary Outcome: CXCL10 in Skin
Description: D-sqaume epidermal discs were used to assess CXCL10 levels from skin.
Time Frame: At time of GVHD diagnosis.
Population: We did not analyze all acute GVHD samples for financial reasons.
Measure: Mean (Standard Error); unit: Skin CXCL10 femtograms/micrograms
Groups:
- Chronic Graft Versus Host Disease: This study arm includes patients who undergo allogeneic hematopoietic cell transplantation at CCHMC and develop chronic graft versus host disease.
Arm/Group | Acute Graft Versus Host Disease | Healthy Controls | Chronic Graft Versus Host Disease
Number analyzed (Participants) | 20 | 10 | 2
Skin CXCL10 femtograms/micrograms | 273 (95) | 41 (76) | 7.5 (2.11)
Statistical Analysis 1: Comparison: Acute Graft Versus Host Disease vs Healthy Controls vs Chronic Graft Versus Host Disease; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Primary Outcome: CXCL10 in Plasma
Description: Plasma was used to assess CXCL10 levels from blood.
Time Frame: At time of GVHD diagnosis.
Population: We did not analyze the plasma collected from patients with chronic skin GVHD; therefore, there is no data to report. We did not analyze all acute GVHD samples for financial reasons.
Measure: Mean (Standard Error); unit: Plasma CXCL10 picograms/microliters
Arm/Group | Acute Graft Versus Host Disease | Healthy Controls
Number analyzed (Participants) | 20 | 10
Plasma CXCL10 picograms/microliters | 5198 (943) | 608 (302)
Statistical Analysis 1: Comparison: Acute Graft Versus Host Disease vs Healthy Controls; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Acute Graft Versus Host Disease | Chronic Graft Versus Host Disease | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/2 | 0/10
Other Adverse Events (participants affected / at risk) | 0/51 | 0/2 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes